CLINICAL TRIAL: NCT02238184
Title: Postmarketing Surveillance Study (as Per §67(6 )AMG [German Drug Law]) of Anticholinergics - Prescribing Pattern and Therapeutic Long Term Value in Patients Suffering From Moderate or Severe Chronic Obstructive Pulmonary Disease
Brief Title: Postmarketing Surveillance Study of Anticholinergics - Prescribing Pattern and Therapeutic Long Term Value in Patients Suffering From Moderate or Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 244.2499
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; oxitropium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Chronic Obstructive Pulmonary Disease: patients receiving Atrovent®
  Interventions: Drug: Atrovent®
- Cronic Obstructive Pulmonary Disease: patients receiving Ventilat®
  Interventions: Drug: Ventilat®

INTERVENTIONS:
Drug: Atrovent®
  Groups: Chronic Obstructive Pulmonary Disease
Drug: Ventilat®
  Groups: Cronic Obstructive Pulmonary Disease

SUMMARY:
To obtain further information on the prescribing pattern and therapeutic long term value in patients suffering from moderate or severs Chronic Obstructive Pulmonary Disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders older than 40 years, who suffer from moderate or severe Chronic Obstructive Pulmonary Disease
* Only patients who showed following diagnosis parameters were to be considered for inclusion

  * FEV1 (Forced expiratory volume in 1 second) and FEV1/VC (vital capacity) <70%
  * Reversibility FEV1 <12% in the last 6 months
  * Smoker or Ex-smoker (>10 Pack years)
  * Asthma to be excluded

Exclusion Criteria:

• Contraindications listed in the Instructions for Use/Summary of Product Characteristics

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive airways disease recruited by registered pneumologists
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2001-01; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Change in overall severity of the clinical picture rated on a 4-point scale | Up to 6 months after first study drug administration
Investigator assessment of improvement of thec linical picture rated on a 6-point symptom profile | Up to 6 months after first study drug administration

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 4-point scale | Up to 6 months after first study drug administration
Assessment of efficacy by patient on a 4-point scale | Up to 6 months after first study drug administration
Assessment of tolerability by investigator on a 4-point scale | Up to 6 months after first study drug administration
Assessment of tolerability by patient on a 4-point scale | Up to 6 months after first study drug administration
Number of patients with adverse drug reactions | Up to 6 months after first study drug administration